CLINICAL TRIAL: NCT07198815
Title: A Preliminary Exploratory Clinical Trial to Evaluate the Efficacy of NPDR-01 Eye Drops in the Treatment of Non-Proliferative Diabetic Retinopathy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLYang
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non-proliferative Diabetic Retinopathy (NPDR); Diabetic Retinal Microangiopathy; Retinal Microaneurysms; Diabetic Retinopathy
Keywords: Diabetic retinopathy; Non-proliferative diabetic retinopathy; Retinal microaneurysms
MeSH Terms: conditions — Microaneurysm; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NPDR-01 Eye Drops Treatment Group (Experimental)
  Interventions: Drug: Investigational Eye Drops (NPDR-01)

INTERVENTIONS:
Drug: Investigational Eye Drops (NPDR-01) — NPDR-01 is an investigational ophthalmic solution administered as one drop (50 μL) to the affected eye(s) once daily for a period of 6 months. It is designed to reduce retinal microaneurysms and slow the progression of non-proliferative diabetic retinopathy.

SUMMARY:
This study aims to explore the preliminary clinical efficacy and safety of NPDR-01 eye drops in patients with non-proliferative diabetic retinopathy (NPDR).

DETAILED DESCRIPTION:
The primary objective is to evaluate the drug's potential to reduce microaneurysm formation, improve retinal lesions, and slow disease progression. The secondary objective is to assess the safety profile of NPDR-01, with a focus on the incidence of ocular adverse events.

ELIGIBILITY:
Inclusion Criteria:

1.1. Patients aged 18 to 75 years diagnosed with type 1 or type 2 diabetes mellitus, with non-proliferative diabetic retinopathy (NPDR) confirmed by a qualified ophthalmologist. NPDR diagnosis must be based on current standard fundus examination or retinal photography and should meet the International Clinical Diabetic Retinopathy Disease Severity Scale, with the presence of microaneurysms.

1.2. Willing and able to comply with study procedures and provide informed consent: Subjects must voluntarily participate in the study, sign the informed consent form, and fully understand the study objectives, potential drug risks, and research procedures. There should be no other ocular diseases causing retinal neovascularization.

1.3. No known significant media opacities that would interfere with fundus image acquisition.

1.4. No history of retinal laser photocoagulation, and no anticipated laser treatment within the next 6 months.

1.5. No history of intravitreal injection therapies, and no anticipated intravitreal treatments within the next 6 months.

1.6. No diabetic macular edema (DME) as defined by central retinal thickness on OCT: <290 μm for females and <305 μm for males (or <305 μm for females and <320 μm for males, depending on the criteria used).

1.7. Clinical fundus examination and ultra-widefield retinal photography show DR changes milder than early proliferative DR (PDR).

1.8. No history of ocular surgery. 1.9. Diabetes history: Duration of diabetes ≥ 1 year; glycemic control with HbA1c ≤ 10%.

1.10. Visual acuity requirement: Best-corrected visual acuity (BCVA) must be better than 20/400, to ensure reliable assessment of drug efficacy.

Exclusion Criteria:

2.1. Age Restrictions: Subjects younger than 35 years or older than 75 years. 2.2. Severe Ocular Complications: Subjects whose diabetic retinopathy has progressed to proliferative diabetic retinopathy (PDR) or who present with clinically significant macular edema (CSME). This includes vitreous hemorrhage, retinal detachment, or other acute complications. Also excluded are subjects with severe optic nerve damage or glaucoma (intraocular pressure > 21 mmHg).

2.3. Poor Diabetes Control: Subjects with HbA1c > 10%, or with highly fluctuating blood glucose levels that may interfere with efficacy evaluation.

2.4. Other Ocular Diseases: Presence of age-related macular degeneration (AMD), retinal vascular occlusion, retinal infections, or other significant ocular pathologies. Also excluded are those with corneal diseases, severe conjunctivitis, or dry eye syndrome that may affect topical ocular drug administration.

2.5. History of Ocular Surgery or Treatments: Subjects who received intraocular injections (e.g., anti-VEGF agents) or retinal laser therapy within the past 6 months. Also excluded are those who recently underwent cataract surgery or other retinal-related surgeries.

2.6. Other Health Conditions: Subjects with abnormal liver function, disorders in ketone body metabolism, or those with serious systemic diseases that may interfere with treatment (e.g., acute heart disease, liver disease, renal failure). History of cancer or current malignancy, or any major illness affecting drug metabolism or immune function.

2.7. Drug Allergy History: Known allergy or hypersensitivity to the study drug or any of its components (e.g., drug carriers, excipients).

2.8. Concomitant Medications: Use of antiplatelet agents (e.g., aspirin, clopidogrel) or anticoagulants (e.g., warfarin, rivaroxaban). Also excluded are those with poorly controlled hypertension, or those who have recently undergone major changes in antihypertensive therapy.

2.9. Pregnant or Lactating Women: Pregnant or breastfeeding women are excluded due to potential drug transmission through the placenta or breast milk that could affect the fetus or infant.

2.10. Other: Subjects who are unwilling or unable to comply with study procedures or follow-up. Any other individuals deemed unsuitable for the study at the discretion of the investigator.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of retinal microaneurysms from baseline to 6 months | Baseline, 1 month, 3 months, and 6 months after treatment initiation
  To evaluate the clinical efficacy of NPDR-01 eye drops in patients with non-proliferative diabetic retinopathy, specifically in reducing the number of retinal microaneurysms, improving retinopathy status, and delaying disease progression.

SECONDARY OUTCOMES:
Incidence of ocular adverse events | Baseline, 1 month, 3 months, and 6 months after treatment initiation